CLINICAL TRIAL: NCT03636061
Title: Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease (The ONSET-1 Study)
Brief Title: Evaluation of the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-002
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OC-01 Low Dose, 0.12 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, Low Dose, 0.12 mg/mL
  Interventions: Drug: OC-01 (varenicline) nasal spray
- OC-01 Mid Dose, 0.6 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray Mid dose, 0.6 mg/mL
  Interventions: Drug: OC-01 (varenicline) nasal spray
- OC-01 High Dose, 1.2 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray High dose, 1.2 mg/mL
  Interventions: Drug: OC-01 (varenicline) nasal spray
- Placebo (Placebo Comparator): Placebo (vehicle) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline) nasal spray — OC-01 (varenicline) nasal spray
  Arms: OC-01 High Dose, 1.2 mg/mL; OC-01 Low Dose, 0.12 mg/mL; OC-01 Mid Dose, 0.6 mg/mL
Drug: Placebo (vehicle) nasal spray — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo on signs and symptoms of dry eye disease

DETAILED DESCRIPTION:
This was a Phase 2b, multicenter, randomized, double-masked, placebo controlled study designed to evaluate the safety and efficacy of OC 01 nasal spray in adult subjects with DED. The study randomized 182 subjects, at least 22 years of age, who had a physician's diagnosis of dry eye disease and met all other study eligibility criteria to receive an application of OC-01 or placebo twice daily (BID) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery within twelve months of Visit 1
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Newport Beach, Newport Beach, California
  - Indianapolis, Indianapolis, Indiana
  - Andover, Andover, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauswirth SG, Kabat AG, Hemphill M, Somaiya K, Hendrix LH, Gibson AA. Safety, adherence and discontinuation in varenicline solution nasal spray clinical trials for dry eye disease. J Comp Eff Res. 2023 Jun;12(6):e220215. doi: 10.57264/cer-2022-0215. Epub 2023 Apr 25. PMID 37096956
- [Derived] Sheppard JD, O'Dell LE, Karpecki PM, Raizman MB, Whitley WO, Blemker G, Hemphill M, Hendrix LH, Gibson A, Macsai M. Does Dry Eye Disease Severity Impact Efficacy of Varenicline Solution Nasal Spray on Sign and Symptom Treatment Outcomes? Optom Vis Sci. 2023 Feb 1;100(2):164-169. doi: 10.1097/OPX.0000000000001986. Epub 2022 Dec 31. PMID 36728653
- [Derived] Nijm LM, Zhu D, Hemphill M, Blemker GL, Hendrix LH, Kabat AG, Gibson AA. Does Menopausal Status Affect Dry Eye Disease Treatment Outcomes with OC-01 (Varenicline Solution) Nasal Spray? A Post Hoc Analysis of ONSET-1 and ONSET-2 Clinical Trials. Ophthalmol Ther. 2023 Feb;12(1):355-364. doi: 10.1007/s40123-022-00607-7. Epub 2022 Nov 18. PMID 36401081
- [Derived] Wirta D, Torkildsen GL, Boehmer B, Hollander DA, Bendert E, Zeng L, Ackermann M, Nau J. ONSET-1 Phase 2b Randomized Trial to Evaluate the Safety and Efficacy of OC-01 (Varenicline Solution) Nasal Spray on Signs and Symptoms of Dry Eye Disease. Cornea. 2022 Oct 1;41(10):1207-1216. doi: 10.1097/ICO.0000000000002941. Epub 2021 Dec 21. PMID 36107843

RESULTS

PARTICIPANT FLOW:
Groups:
- OC-01 Low Dose, 0.12 mg/ml: OC-01 0.12 mg/ml nasal spray BID for 28 days
- OC-01 Mid Dose, 0.6 mg/ml: OC-01 0.6 mg/ml nasal spray BID for 28 days
- OC-01 High Dose, 1.2 mg/ml: OC-01 1.2 mg/ml nasal spray BID for 28 days
Period: Overall Study
Arm/Group | OC-01 Low Dose, 0.12 mg/ml | OC-01 Mid Dose, 0.6 mg/ml | OC-01 High Dose, 1.2 mg/ml | Placebo
Started | 47 | 48 | 44 | 43
Completed | 47 | 46 | 40 | 43
Not Completed | 0 | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Vehicle nasal spray
- Total: Total of all reporting groups
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 44 | 43 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (12.7) | 66.5 (9.4) | 67.4 (10.6) | 64 (10.3) | 65.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 35 | 32 | 137
  Male | 11 | 14 | 9 | 11 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 2 | 5 | 18
  Not Hispanic or Latino | 39 | 45 | 42 | 38 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 3 | 4 | 0 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 4 | 6 | 2 | 14
  White | 42 | 39 | 36 | 40 | 157
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 44 | 43 | 182
Schirmer's Test Score [Mean (Standard Deviation); unit: mm] — Schirmer's test score from 0-35 mm where a higher score is indicative of a better outcome.
  mm | 5.2 (3.1) | 4.8 (2.7) | 5.5 (3.0) | 4.5 (2.9) | 5.0 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Schirmer's Test Score From Baseline to 28 Days
Description: The primary end point was the change in anesthetized Schirmer's Test Score (STS) from baseline to 28 days in the study eye following treatment with OC-01. Schirmer's test score from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: 28 Days [Visit 1 (baseline) and Visit 5 (28 days)]
Population: Subjects in ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: score on a scale, mm
Groups:
- OC-01 Low Dose, 0.12 mg/mL: OC-01 0.12 mg/ml nasal spray
- OC-01 Mid Dose, 0.6 mg/ML: OC-01 0.6 mg/ml nasal spray
- OC-01 High Dose, 1.2 mg/mL: OC-01 1.2 mg/ml nasal spray
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/ML | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 47 | 46 | 40 | 43
score on a scale, mm | 10.1 (1.26) | 11.7 (1.27) | 11.0 (1.39) | 3.2 (1.31)

2. Secondary Outcome: Change From Baseline in Eye Dryness Score From Baseline to Day 28
Description: Change in Eye Dryness Score from baseline to 28 days. Eye Dryness (EDS) on a Visual Analogue Scale (VAS) from 0 (no discomfort) to 100 (maximum discomfort) millimeters where a lower score is indicative of a better outcome.
Time Frame: 28 days [Visit 1 (baseline and Visit 5 (28 days)]
Population: Subjects in the ITT-LOCF population. The overall number of participants is different because these outcomes were assessed ar different visits 7 days apart and some subjects were not able to attend the Day 21 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale, mm
Arm/Group | OC-01 Low Dose, 0.12 mg/ml | OC-01 Mid Dose, 0.6 mg/ml | OC-01 High Dose, 1.2 mg/ml | Placebo
Number analyzed (Participants) | 47 | 46 | 40 | 43
score on a scale, mm | -11.6 (3.63) | -18.9 (3.67) | -15.6 (4.02) | -5.4 (3.8)

3. Secondary Outcome: Change From Baseline to Day 21 in Eye Dryness Score at 5 Minutes Post Treatment in the CAE.
Description: Change from baseline to Day 21 in Eye Dryness Score at 5 minutes post treatment in the CAE. Eye Dryness (EDS) on a Visual Analogue Scale (VAS) from 0 (no discomfort) to 100 (maximum discomfort) millimeters where a lower score is indicative of a better outcome.
Time Frame: 21 days [Visit 1 (baseline) and Visit 4 (21 days)]
Population: Subjects in the ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale, mm
Arm/Group | OC-01 Low Dose, 0.12 mg/ml | OC-01 Mid Dose, 0.6 mg/ml | OC-01 High Dose, 1.2 mg/ml | Placebo
Number analyzed (Participants) | 44 | 45 | 38 | 42
score on a scale, mm | -8.1 (2.7) | -16.0 (2.7) | -18.4 (3.0) | -4.4 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug administration until the final study visit at Visit 5 (28 days)
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/48 | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 33/47 | 44/48 | 41/44 | 11/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC-01 Low Dose, 0.12 mg/mL (N=47) | OC-01 Mid Dose, 0.6 mg/mL (N=48) | OC-01 High Dose, 1.2 mg/mL (N=44) | Placebo (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC-01 Low Dose, 0.12 mg/mL (N=47) | OC-01 Mid Dose, 0.6 mg/mL (N=48) | OC-01 High Dose, 1.2 mg/mL (N=44) | Placebo (N=43)
Ocular TEAEs (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 7 (7)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival deposit (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairement (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 38 (38) | 37 (37) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 11 (11) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 9 (9) | 0 (0)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 3 (3) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Instillation site irritation (General disorders) | 3 (3) | 8 (8) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03636061/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03636061/SAP_003.pdf